CLINICAL TRIAL: NCT06959264
Title: Effect of Virtual Reality Goggles on Anxiety, Comfort and Complications in Patients Undergoing Transrectal Ultrasound-guided Prostate Biopsy: A Randomised Controlled Study
Brief Title: Effect of Virtual Reality Goggles on Anxiety, Comfort and Complications in Patients Undergoing Transrectal Ultrasound-guided Prostate Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tarsus University (Other)
Collaborators: Mersin University (Other)
Responsible Party: Principal Investigator, Gamze BOZKUL, Dr, Tarsus University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: TU-BOZKUL-012
Record Dates: First submitted 2025-04-26; First posted 2025-05-06 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Prostate Biopsy
Keywords: Virtual Reality; Anxiety; Comfort; Complication; Nursing; Prostate biopsy
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: During the data collection process, when the patients come to the urology outpatient clinic, their inclusion status will be evaluated by the researcher M.B. A total of 70 patients in the sample group determined by randomization will be divided into A and B groups created by the same statistician in the computer environment by block randomization (1:1 ratio) method according to the order of arrival. The A and B status of the study or control group will be determined by coin toss at the beginning of the study. The information showing that the patients included in the research sample are assigned to group A and B according to the randomization table will be placed in an opaque envelope. This envelope will be kept by the researcher (GAU) and when the researchers (GB and EKD) go to the patient for the application, they will open the envelope after filling out the "Informed Consent Form" and learn which group the patient is in. While the researchers (GB and EKD) will be blinded in the assign
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality group (Experimental): Patients in the study group will be shown a video with virtual reality glasses during the procedure. Patients will be asked to wear a virtual reality goggles (VR Shinecon G12 3d Virtual Reality Goggles Black 4.5-7.0 Inch) compatible with a mobile phone (Xiaomi Redmi Note 8 Pro 2019 model) with android operating system in supine position and minimizing sound loss. With the virtual reality goggles, nature landscapes with a relaxing music background will be watched by adjusting the volume at the level desired by the patient. Virtual reality goggles will be applied during the procedure.
  Interventions: Other: Virtual reality
- Control group (No Intervention): The control group will not receive any intervention.

INTERVENTIONS:
Other: Virtual reality — Patients in the study group will be shown a video with virtual reality glasses during the procedure. Patients will be asked to wear a virtual reality goggles (VR Shinecon G12 3d Virtual Reality Goggles Black 4.5-7.0 Inch) compatible with a mobile phone (Xiaomi Redmi Note 8 Pro 2019 model) with android operating system in supine position and minimizing sound loss. With the virtual reality goggles, nature landscapes with a relaxing music background will be watched by adjusting the volume at the level desired by the patient. Virtual reality goggles will be applied during the urodynamic procedure.
  Arms: Virtual reality group

SUMMARY:
This study was aimed to determine the effect of virtual reality goggles on anxiety, comfort and complication development in patients undergoing transrectal ultrasound-guided prostate biopsy in a randomized controlled experimental study. The study will be conducted with individuals who applied to the Department of Urology of Mersin University Hospital. The minimum sample calculation with 95% power was calculated as a total of 70, 35 in each group, in the G*Power (3.1) program. Introductory Information Form, State Anxiety Scale, Complication Follow-up Form and Visual Analog Scale will be used to collect the data. Introductory Information Form, State Anxiety Scale and Visual Analog Scale will be filled in the patients. After the forms are applied to the patients and recorded, it will be determined whether they will be in the study or control group according to the randomization schedule. Patients in the study group will be shown a video with virtual reality glasses during the procedure. Virtual reality goggles will be used to watch nature landscapes with relaxing music background, adjusted at the level of volume desired by the patient. Virtual reality goggles will be applied during the procedure. The control group will not receive any intervention. After the virtual reality application, anxiety levels and comfort levels will be re-evaluated after the procedure. The patients will be called by the researchers after 24 hours and the Complication Follow-up Form will be filled out. The data obtained in the study will be analyzed using SPSS (Statistical Package for Social Sciences) for Windows 25.0 program.

DETAILED DESCRIPTION:
This study was aimed to determine the effect of virtual reality goggles on anxiety, comfort and complication development in patients undergoing transrectal ultrasound-guided prostate biopsy in a randomized controlled experimental study. The study will be conducted with individuals who applied to the Department of Urology of Mersin University Hospital between May 2025 and May 2026 and met the sampling criteria. Taking the effect size 0.87 as a reference, d=0.87, (1- α, bidirectional), the minimum sample calculation with 95% power was calculated as a total of 70, 35 in each group, in the G*Power (3.1) program. Introductory Information Form, State Anxiety Scale, Complication Follow-up Form and Visual Analog Scale will be used to collect the data. Introductory Information Form, State Anxiety Scale and Visual Analog Scale will be filled in the patients. After the forms are applied to the patients and recorded, it will be determined whether they will be in the study or control group according to the randomization schedule. Patients in the study group will be shown a video with virtual reality glasses during the procedure. Patients will be asked to wear a virtual reality goggles (VR Shinecon G12 3d Virtual Reality Goggles Black 4.5-7.0 Inch) compatible with a mobile phone (Xiaomi Redmi Note 8 Pro 2019 model) with android operating system and minimizing sound loss in the supine position.Virtual reality goggles will be used to watch nature landscapes with relaxing music background, adjusted at the level of volume desired by the patient. Virtual reality goggles will be applied during the procedure. The control group will not receive any intervention. After the virtual reality application, anxiety levels and comfort levels will be re-evaluated after the procedure. The patients will be called by the researchers after 24 hours and the Complication Follow-up Form will be filled out. The data obtained in the study will be analyzed using SPSS (Statistical Package for Social Sciences) for Windows 25.0 program.

ELIGIBILITY:
Inclusion Criteria:

* Who agreed to participate in the study,
* Patients over 18 years of age
* Conscious, oriented and cooperative,
* No communication problems,
* Transrectal ultrasound guided prostate biopsy procedure,
* No physical problems that would prevent the application of virtual reality goggles,
* No previous experience with virtual reality glasses,
* Undiagnosed anxiety,
* No medication for anxiety
* Patients without mental disorders

Exclusion Criteria:

* Who did not agree to participate in the study,

  * Patients under 18 years of age,
  * Conscious, oriented and uncooperative,
  * Communication problems,
  * No transrectal ultrasound-guided prostate biopsy procedure,
  * With a physical problem that would prevent the application of virtual reality goggles,
  * Diagnosed with anxiety,
  * Taking medication for anxiety (anxiolytics, antidepressants, antipsychotics, etc.),
  * Patients with mental disorders

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The procedure is specific for men because it is a prostate biopsy
Enrollment: 70 (Actual)
Dates: Start 2025-04-28 (Actual); Primary Completion 2025-12-15 (Actual); Study Completion 2025-12-15 (Actual)

PRIMARY OUTCOMES:
Anxiety | 6 months
  The State Anxiety Scale : In this study, the DAQ, which is structured to measure momentary feelings, was used. Its Turkish validity and reliability was conducted by Öner and Le Compte in 1983. The DAQ consists of 20 questions on a four-point Likert scale. The statements in the DAQ are evaluated as not at all (1), a little (2), a lot (3) and completely (4). In this section, the statements are divided into direct and reversed statements. Inverted statements: 1st, 2nd, 5th, 5th, 8th, 8th, 10th, 11th, 15th, 16th, 19th, 20th items. The total score of the reversed statements is subtracted from the total score of the direct statements and the number 50, which is the invariant value of the DAQ, is added to the value obtained and the DAQ score is calculated. The scale score ranges between 20-80 and an increase in the score indicates an increase in the level of anxiety.
Comfort | 6 months
  Visual Analog Scale: It is a scale that provides a subjective assessment of comfort on a horizontal or vertical line from 0 -10 to evaluate the level of comfort.
Complications | 6 months
  Patients will be questioned about bleeding in the first urine, hematuria, hematospermia, rectal bleeding, anal pain, dysuria and urinary retention within 24 hours after the procedure and recorded on the form.

CONTACTS AND LOCATIONS:
Overall Officials: Gülay Altun Uğraş, Principal Investigator — Mersin University; MURAT Bozlu, Principal Investigator — Mersin University
Locations (1):
- Tarsus University, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Thomson A, Li M, Grummet J, Sengupta S. Transperineal prostate biopsy: a review of technique. Transl Androl Urol. 2020 Dec;9(6):3009-3017. doi: 10.21037/tau.2019.12.40. PMID 33457274
- [Result] Genc H, Korkmaz M, Akkurt A. The Effect of Virtual Reality Glasses and Stress Balls on Pain and Vital Findings During Transrectal Prostate Biopsy: A Randomized Controlled Trial. J Perianesth Nurs. 2022 Jun;37(3):344-350. doi: 10.1016/j.jopan.2021.09.006. Epub 2022 Apr 7. PMID 35397973